CLINICAL TRIAL: NCT07031804
Title: Expectation Effects on Emotional Processing
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Stefanie Brassen, Prof. Dr., Universitätsklinikum Hamburg-Eppendorf
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Exface
Record Dates: First submitted 2025-06-04; First posted 2025-06-22 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Expectation Effects on Emotional Processing
Keywords: Positive expectation; Treatment expectation; fMRI; Emotional processing; Placebo

STUDY DESIGN:
Intervention Model Description: A cross-over design will be employed by giving a saline nasal spray introduced either as oxytocin or as saline.
Who Masked: Participant
Masking Description: Participants will be blinded to the real substance (saline nasal spray).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo - Control (Experimental): Participants in this group receive sham oxytocin on the first study day.
  Interventions: Other: Saline Nasal Spray
- Control - Placebo (Experimental): Participants in this group receive sham oxytocin on the second study day
  Interventions: Other: Saline Nasal Spray

INTERVENTIONS:
Other: Saline Nasal Spray — A saline nasal spray will be introduced as saline on the first day (no induced expectations) and as oxytocin on the second day (induced positive expectations)
  Arms: Control - Placebo
Other: Saline Nasal Spray — A saline nasal spray will be introduced as oxytocin on the first day (induced positive expectations) and as saline on the second day (no induced positive expectations)
  Arms: Placebo - Control

SUMMARY:
Understanding the mechanisms underlying expectation effects in the affective domain can provide valuable insights into possible therapeutic interventions for mood disorders. Studies have consistently found that expectations can influence emotional experiences. Recently, it has been shown that top-down cognitive control is critical in inducing instruction-based affective placebo effects. However, changes in the emotional system over time not only rely on higher-level cognitive processes but also on more automatic mechanisms shaped by learning and past experiences. How such mechanisms are involved in affective placebo effects is relatively unknown, but is particularly interesting in light of findings showing that previous experiences of successful treatments are an important determinant of placebo responses.

This study aims to investigate the neurobehavioral mechanisms of how expectations and prior experiences modulate emotional processing. Healthy adults (N = 51, 50% women) will be recruited to participate in a cross-over fMRI study involving two conditions: positive expectation induction (placebo) and a control condition with no induced expectations. Participants will perform an emotion classification task under each condition. The investigators hypothesize that positive expectations enhance mood and improve the accuracy of recognizing happy facial expressions. Further, they hypothesize that affective expectations are represented in fMRI signal patterns in networks involved in face perception, emotional processing, and cognitive control.

DETAILED DESCRIPTION:
Background:

Research demonstrated that positive expectations are related to a perception bias towards positive information and changes in neural networks of affective processing. However, it's unclear how underlying expectancy effects modulate response biases to emotional inputs. A recent study showed the importance of cognitive control and top-down regulation in expectation effects on emotional processing, mechanisms that may be less effective in cognitively vulnerable individuals, such as those with depression. Research on placebo analgesia indicates that not only such higher level-processes but also lower-level processes play a significant role in placebo effects. How such lower level processes are involved in affective placebo effects is relatively unknown but would be highly relevant given that long-term modulation of the emotional system also relies on computationally less costly bottom-up processes typically shaped by learning and experiences. Therefore, this study aims to investigate the neurobehavioral mechanisms of how expectations and prior experiences modulate emotional processing.

Recruitment plan:

Healthy participants will be recruited through an online advertisement on a voluntary basis. An initial short screening to assess basic eligibility (see inclusion and exclusion criteria) will take place over the phone, followed by an extensive screening on site, including the following questionnaires:

* Demographics
* Education
* Generic rating scale for previous treatment experiences, treatment expectations, and treatment effects (G-EEE)
* Beck Depression Inventory (BDI)

Design:

The study consists of three days: one screening day and two study days. On the screening day, in addition to assessing eligibility, participants will receive a saline nasal spray that is introduced as oxytocin. Treatment expectations will be induced via an established expectation induction protocol that systematically manipulates expectations in the context of face perception. Positive expectations about "oxytocin" will be induced via a video documentary detailing the mechanisms of oxytocin, highlighting its mood-enhancing effects and role in emotional processing. In detail, participants will complete a short training of an emotion classification task, view the video documentary, self-administer the nasal spray, rate their expectations using a visual analogue scale (VAS, from "no expected mood enhancement" to "strong expected mood enhancement"), and then complete the same training again. However, the second training is covertly manipulated and is designed to facilitate the detection of happy facial expressions. At the end of the day they will rate their experience with a VAS (from "experienced no positive mood change" to "experienced a large positive mood change"). This expectation induction combined with the covertly manipulated training is already implemented on the screening day to establish positive prior experiences associated with "oxytocin" and therefore enhance placebo effects on the study days. If a participant does not believe in the treatment on the screening day, they will not be included for the main study.

In a cross-over experiment, on two study days that are one week apart, participants will undergo fMRI scanning. Before scanning, participants will receive a saline nasal spray that is either introduced as oxytocin (placebo condition) or saline (control condition) in a counter-balanced design. Expectations will be reinforced via the video documentary. After the video, participants will receive verbal instructions about their assigned condition for that day (either "oxytocin" or control), self-administer the nasal spray, and rate their expectations. Depending on the assigned condition, participants will then either complete a standard training (control condition) or a covertly manipulated training ("oxytocin" condition). Participants will assess their current mood (using a VAS) at three time points: before nasal spray administration, after the manipulated training and after the fMRI scan. At the end of each study day, participants will rate their experience. While in the scanner, an emotion classification task is performed, in which participants label images of subtle emotional face expressions, varying in emotional intensity, as happy, fearful, or neutral. As a control measure, horizontal gaze trajectories (fixation and gaze shifts patterns) will be recorded using eye-tracking.

Hypotheses:

The investigators will examine the effects of positive expectations on mood state and task accuracy and investigate how positive expectations modulate uni- and multivariate fMRI signal patterns associated with the processing and categorization of emotional stimuli. More specifically, they hypothesize the following:

* Positive expectations enhance mood and improve the accuracy of detecting subtle happy facial expressions.
* fMRI patterns in sensory, affective, and cognitive areas in response to subtle happy faces are more similar to patterns evoked by unambiguous happy face localizers in the positive treatment expectation condition.
* Pattern dissimilarity across happiness intensities decreases in the placebo condition.
* Expectation effects on mood, happy face accuracy, and neural patterns are related to expectation ratings and measures of prior experience induced by the manipulated training.

Analysis plan:

For the behavioral analysis, statistical protocols developed in our lab will be applied, with a main focus on response threshold and sensitivity derived from psychometric functions. The effects of expectation on mood state and task accuracy and post-treatment experience will be assessed using statistical tests from the general linear model framework, including t-tests, repeated measures ANOVA and Pearson correlations. Statistical significance will be assumed based on an alpha value of 0.05. Emotion-specific psychometric response functions will be derived from regressing individual accuracy rates from the placebo condition on the control condition. The psychometric response functions will allow us to disentangle expectation effects with respect to response tendencies (intercept) and perceptual sensitivity (slope).

For the univariate fMRI analysis, a two-level random effects general linear model (GLM) approach will be employed, modeling task-related activity using the hemodynamic response function (HRF). Whole-brain analysis (cluster-level corrected) and a small-volume regions of interest (ROI) approach will be applied (p < .05 FWE corrected). A multivariate representational similarity analysis (RSA) approach will be used to compare the similarity of fMRI patterns during subtle emotional face presentation with patterns derived from unambiguous emotional face localizers. RSA protocols have previously been developed in our lab.

The here presented study is part of the collaborative research center (CRC) SFB/TRR289 and is funded by the Deutsche Forschungsgemeinschaft (DFG, ID: 422744262).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-35 years
* MRI compatible
* Medical information and signed declaration of consent
* Normal or corrected to normal vision
* German speaking

Exclusion Criteria:

* No informed consent
* Current intake of central nervous system active drugs
* Under influence of alcohol
* BDI score above 12
* Significant acute somatic or neurological diseases
* History of psychiatric or neurological disorders
* Pregnancy/ breastfeeding
* Acute nasal diseases or injuries
* MR-specific exclusion criteria (claustrophobia, pacemaker, non-MR compatible metallic objects)
* fMRI data with strong artefacts or excessive movement will be excluded from analysis
* If a participant does not believe in the treatment on the screening day, they will not be included for the main study days
* If a participant drops out after study day one, they will be excluded from the analysis

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Effects of positive expectation on mood | On both day 1 and day 2, measurements will be taken before the intervention (VAS baseline), 5 minutes after nasal spray application, and after the scanning (~ 60 minutes after nasal spray application).
  Mood ratings via visual analogue scale (VAS), consisting of a scale from 0 to 200 points (0 meaning unhappy; 200 meaning happy). VAS will be extracted as a raw score and then normalized to the baseline VAS. It will be analyzed to assess differences between interventions (placebo and control) and to evaluate changes over time throughout the experiment.
Effects of positive expectation on task performance data | Approximately 15 minutes after the nasal spray application, participants will perform an emotion classification task for 40 minutes while lying in the scanner on each day.
  Accuracies from the emotion classification task will be extracted and sampled for 3 emotional (happy, fearful and neutral) conditions for both interventions (Placebo and Control). Performance during the placebo condition will be regressed onto performance during the control condition for each emotion. The resulting emotion-specific psychometric response functions will allow us to disentangle expectation effects with respect to response tendencies (the intercept) and discrimination ability (the slope).
Effects of positive expectation on blood oxygen level dependent (BOLD) signals | Approximately 15 minutes after the nasal spray application, participants will lie in the scanner for ~ 40 minutes while performing the emotion classification task on each day.
  Functional magnetic resonance imaging will be used to extract and analyze BOLD signals (regions of interest and whole brain) in response to the emotional conditions and interventions. Univariate and multivariate analyses will be performed to compare activation profiles and the similarity of fMRI patterns during placebo and control.

CONTACTS AND LOCATIONS:
Overall Officials: Stefanie Brassen, Prof. Dr., Principal Investigator — Department of Systems Neuroscience, University Hospital Hamburg-Eppendorf, Hamburg, Germany
Locations (1):
- University Medical Center Hamburg-Eppendorf, Institute of Systems Neuroscience, Hamburg, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: With Publication

REFERENCES:
- [Background] Mostauli A, Rauh J, Gamer M, Buchel C, Rief W, Brassen S. Placebo treatment entails resource-dependent downregulation of negative inputs. Sci Rep. 2025 Mar 17;15(1):9088. doi: 10.1038/s41598-025-93589-y. PMID 40097556
- [Background] Baker J, Gamer M, Rauh J, Brassen S. Placebo induced expectations of mood enhancement generate a positivity effect in emotional processing. Sci Rep. 2022 Mar 29;12(1):5345. doi: 10.1038/s41598-022-09342-2. PMID 35351936